CLINICAL TRIAL: NCT03322176
Title: Medical Provider Experience Assessment Healthcare Decisions Post-Testing, Risk-Reducing, and Preventative Strategies Using LYNCH Genetic Testing
Brief Title: Healthcare Decisions Post-Testing, Risk-reducing and Preventative Strategies Using LYNCH Genetic Testing Reducing, and Preventative Strategies Using LYNCH Genetic Testing
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Data Collection Analysis Business Management (Other)
Collaborators: PAS Research Services (Other)
Responsible Party: Sponsor
Other Study IDs: PAS1461
Record Dates: First submitted 2017-10-24; First posted 2017-10-26 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Colon Cancer; Endometrial Cancer
MeSH Terms: conditions — Colonic Neoplasms; Endometrial Neoplasms | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Genetic testing — LYNCH genetic testing

SUMMARY:
Increase surveillance for LYNCH Syndrome

DETAILED DESCRIPTION:
The purpose of this minimal risk, observational survey is to increase surveillance for Lynch Syndrome (hereditary non-polyposis colon cancer), Colorectal, and Endometrial cancer, also to determine targeted risk-reducing and preventative strategies.

ELIGIBILITY:
Inclusion Criteria:

* Must be a Medical Practitioner

  * Medical Doctor (MD)
  * Doctor of Osteopathic (DO)
  * Physician Assistant (PA)
  * Advanced Practice Registered Nurse (APRN)
  * Nurse Practitioner (NP)
* Must have a current standard operating procedure that includes obtaining/reviewing medical history and family medical history.

Exclusion Criteria:

* Government-funded insurance data cannot be included in the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: collecting data and reviewing the Principal Investigators' (P.I.) Standard Operating Procedures (SOP) on Lynch genetic testing and changes made to their specific SOP.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-10-17 (Actual); Primary Completion 2020-10-17 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Provider Structures and Processes | 36 months
  Plan of Care Changes due to LYNCH genetic testing. Provider based observational survey system on the health and well-being of patients and populations

CONTACTS AND LOCATIONS:
Locations (1):
- DCABM, Land O' Lakes, Florida, United States

IPD SHARING:
Plan to Share IPD: No